CLINICAL TRIAL: NCT01407692
Title: Effect of Menstrual Cycle Hormone Changes on Eating Behavior and Nutrient Metabolism
Brief Title: Menstrual Cycle Hormones and Eating Behavior
Acronym: FL-84
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: WHNRC 221594-1
Record Dates: First submitted 2011-07-26; First posted 2011-08-02 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Dietary Habits; Food Preference
Keywords: menstrual cycle; estrogen
MeSH Terms: conditions — Feeding Behavior; Food Preferences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine samples may be retained for future testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the phase of the menstrual cycle (opposed versus unopposed estrogen phase) affects eating behavior, including types of foods preferred, wanting/desire for specific foods, and perception of hunger.

DETAILED DESCRIPTION:
This is an observational study to investigate the effect of endogenous estrogen (E2) and progesterone (P4) levels on eating behavior and energy-yielding nutrient metabolism. Eating behavior will be assessed during a complete menstrual cycle during the first month of the study. Participants will track the follicular and luteal phases of their menstrual cycle using urinary leuteinizing hormone (LH) kits, they will record information about their food intake, eating behaviors, and appetite in their home environments, and they will complete two laboratory test days: one test day scheduled during their follicular phase, and one test day scheduled during their luteal phase.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 20-30 Kg/m2
* regular menstrual cycles
* sedentary lifestyle (physical activity not more than 30 minutes per day three times a week)

Exclusion Criteria:

* Fasting blood sugar greater than 110 mg/dL
* Systolic Blood Pressure greater than 140 mmHg
* Diastolic Blood Pressure greater than 90 mmHg
* Fasting triglycerides greater than 120 mg/dL
* Documented or self-reported chronic disorders such as arthritis, or other inflammatory diseases
* Women who are Post-menopausal or Peri-menopausal
* Pre-menopausal women who are pregnant, uni/multiparous, taking oral contraceptives, or who have menstrual cycles lasting less than 20 days or greater than 45 days, polycystic ovary syndrome (PCOS), amenorrhea, eumenorrhoea, or polymenorrhoea.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, premenopausal women.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Eating behavior | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  Eating behavior, including types of foods preferred, wanting/desire for specific foods, and perception of hunger will be measured using four questionnaires; Eating inventory: to assess dietary restraint, Stanford Brief Physical Activity Questionnaire, Food craving questionnaire, Eating behavior and attitudes questionnaire

SECONDARY OUTCOMES:
Insulin sensitivity | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  To determine if the phase of the menstrual cycle affects insulin sensitivity, we will measure plasma insulin, glucose and non-esterified fatty acids (NEFA).
Serum lipid profile changes | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  Blood samples will be analyzed for lipids and lipoproteins, including apoproteins A1, B, C-II, C-III, and E.
Urinary c-peptide | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  The level of urinary C-peptide and creatinine will be measured in a 24-hour urine collection.
Estradiol | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  Estradiol measured in serum in relation to appetite variables
progesterone | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  Progesterone measured in serum in relation to appetite variables
Dehydroepiandrosterone (DHEA) | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  Dehydroepiandrosterone measured in serum in relation to appetite variables
Sex Hormone Binding Globulin (SHBG) | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  SHBG measured in serum in relation to appetite variables
Endocannabinoid profile | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  Endocannabinoid profile measured in serum to assess appetite
Leptin | At follicular (day 11) and luteal (day 26) phase of menstrual cycle
  Leptin measured in serum to assess appetite

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Keim, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Derived] Krishnan S, Agrawal K, Tryon RR, Welch LC, Horn WF, Newman JW, Keim NL. Structural equation modeling of food craving across the menstrual cycle using behavioral, neuroendocrine, and metabolic factors. Physiol Behav. 2018 Oct 15;195:28-36. doi: 10.1016/j.physbeh.2018.07.011. Epub 2018 Jul 18. PMID 30031087
- [Derived] Krishnan S, Tryon RR, Horn WF, Welch L, Keim NL. Estradiol, SHBG and leptin interplay with food craving and intake across the menstrual cycle. Physiol Behav. 2016 Oct 15;165:304-12. doi: 10.1016/j.physbeh.2016.08.010. Epub 2016 Aug 12. PMID 27527001
- See also: United States Department of Agriculture, ARS, Western Human Nutrition Research Center — https://www.ars.usda.gov/pacific-west-area/davis-ca/whnrc/